CLINICAL TRIAL: NCT00355160
Title: Non-Rhinologic Etiologies of Headaches and Facial Pain in Tertiary Care Setting
Status: Completed | Type: Observational
Sponsor: Penn State University (Other)
Responsible Party: Principal Investigator, Johnathan McGinn, Associate Professor, Penn State University
Other Study IDs: 23218EP
Record Dates: First submitted 2006-07-19; First posted 2006-07-21 (Estimated); Last update posted 2013-05-15 (Estimated); Status verified 2013-05

CONDITIONS: Headache; Sinusitis; Rhinitis; Facial Pain
Keywords: Headache; Sinusitis; Rhinitis; Facial Pain
MeSH Terms: conditions — Headache; Sinusitis; Rhinitis; Facial Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The study serves to investigate the type and prevalence of non-rhinologic headaches seen through a academic otolaryngology practice.The study encompasses survey questionnaires, review of CT images, and physical examination/nasal endoscopy findings.

DETAILED DESCRIPTION:
1. Rationale Our aim is to conduct a prospective study to assess the patients referred for rhinosinusitis to a tertiary rhinologic practice whose symptoms include headache/facial pain, but have no evidence of significant rhinologic disease and determine whether a neurologic etiology is responsible for headaches or facial pressure/pain symptoms.
2. Key Objectives 1. Assess prevalence of headache syndromes in patients with primary complaints of facial pain and headaches. 2. Correlate average Lund McKay CT scan score in patients with headache syndromes
3. Study Population Patients referred to Dr. McGinn's otorhinolaryngologic practice for assessment of rhinosinusitis who do not meet the criteria for the diagnosis of rhinosinusitis.
4. Major Inclusion & Exclusion Criteria Inclusion criteria include patients greater than 18 years of age, literate in the English language, referred by a physician for primary complaint of "sinusitis", major symptomatic complaint of headache or facial pain/pressure, CT scan must have been performed prior and available for review at the time of visit. Exclusion criteria include evidence of chronic rhinosinusitis, a modified LM score greater than 2, pregnancy, history of prior facial trauma or tumor in the head and neck region, specifically the nasal area, past history of autoimmune disorder affecting the head and neck region (e.g., Wegener's granulomatosis).
5. Allocation to Groups None
6. Procedures: Participants will be asked to complete a headache questionnaire and the SNOT-20 questionnaire (a validated tool developed by Dr. Picirillo). Information from the subjects' medical records related to their headaches and facial pain will be recorded for the research. This information will include the results of the CT scan, nasal endoscopic exam, and clinical exam.
7. Major Risks and Discomforts: Loss of confidentiality.
8. Confidentiality: No patient names or other identifying information will be revealed in the course of the study. There will be no direct patient identifiers on the database utilized for this study. The initial patient form scanned into the database will utilize a coded identifier based on chronological order in order to prevent inadvertent disclosure of private medical data. The code will be kept secure in a locked filing cabinet in the principal investigator's office and destroyed once the data are collected and the study is completed.
9. Investigator Qualifications & Specific Roles in the Research Johnathan M. McGinn, MD is a board certified otolaryngologist.
10. Study Site Location(s) - Hershey Medical Center outpatient clinic

ELIGIBILITY:
Inclusion Criteria:

* patients greater than 18 years of age
* literate in the English language
* referred by a physician for primary complaint of "sinusitis"
* major symptomatic complaint of headache or facial pain/pressure
* CT scan must have been performed prior and available for review at the time of visit

Exclusion Criteria:

* evidence of chronic rhinosinusitis
* a modified Lund Mackay score greater than 2 on CT
* pregnancy
* history of prior facial trauma or tumor in the head and neck region, specifically the nasal area
* past history of autoimmune disorder affecting the head and neck region (e.g., Wegener's granulomatosis).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pateints presenting to our clinic with a diagnosis of "sinusitis" by referring physicians with facial pain and/or headache as key complaint, ut who have no clincal evidence of sinusitis by CT scan or examination
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2006-07; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Headache subtype | completion of questionnaire
  Questionnaire study - headache subtype determined by data provided. No clinical intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Johnathan D McGinn, MD, Principal Investigator — Penn State College of Medicine, Penn State Milton S. Hershey Medical Center
Locations (1):
- Penn State College of Medicine, Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

REFERENCES:
- See also: Related Info — http://www.hmc.psu.edu/otolaryngology/